CLINICAL TRIAL: NCT05794243
Title: An Open-Label, Multiple-Dose Study to Investigate the Pharmacokinetics of LY3493269 Oral Formulations Administered in a Fed or Fasted State in Healthy Participants
Brief Title: A Multiple-Dose Study of LY3493269 in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Following preplanned review of the safety and pharmacokinetic data from Part A, it was determined that sufficient data had been obtained. The decision was made to not proceed with Part B and the study was terminated early.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18360; J1X-MC-GZHI (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Healthy
MeSH Terms: interventions — decanoic acid; Neprilysin; N-(8-(2-hydroxybenzoyl)amino)caprylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A: 4 mg LY3493269 Test Capsule 1 + 280 mg C10 (Fasted) (Experimental): * Participants were administered oral doses of 4 milligram (mg) LY3493269 test capsule formulation 1, co-administered with 280 mg of sodium caprate (C10).
  * This regimen was administered once daily on Days 1, 2, and 3, following an overnight fast.
  Interventions: Drug: LY3493269; Drug: Sodium Caprate (C10)
- Part A: 4 mg LY3493269 Test Capsule 2 + 280 mg C10 (Fasted) (Experimental): * Participants were administered oral doses of 4 mg LY3493269 test capsule formulation 2, co-administered with 280 mg of C10.
  * This regimen was administered once daily on Days 1, 2, and 3, following an overnight fast.
  Interventions: Drug: LY3493269; Drug: Sodium Caprate (C10)
- Part A: 4 mg LY3493269 Reference Tablet + 300 mg SNAC (Fasted) (Experimental): * Participants were administered oral doses of 4 mg LY3493269 reference tablet formulation, co-administered with 300 mg of salcaprozate sodium (SNAC).
  * This regimen was administered once daily on Days 1, 2, and 3, following an overnight fast.
  Interventions: Drug: LY3493269; Drug: Salcaprozate Sodium (SNAC)
- Part B: LY3493269 (Experimental): The formulation of the LY3493269 test capsule (1,2) or reference tablet were planned to be determined based on the initial review of safety and pharmacokinetic data from Part A.
  Interventions: Drug: LY3493269

INTERVENTIONS:
Drug: LY3493269 — Administered orally.
Drug: Sodium Caprate (C10) — Administered orally.
  Arms: Part A: 4 mg LY3493269 Test Capsule 1 + 280 mg C10 (Fasted); Part A: 4 mg LY3493269 Test Capsule 2 + 280 mg C10 (Fasted)
Drug: Salcaprozate Sodium (SNAC) — Administered orally.
  Arms: Part A: 4 mg LY3493269 Reference Tablet + 300 mg SNAC (Fasted)

SUMMARY:
The main purpose of this study is to conduct blood tests to measure how much LY3493269 is in the bloodstream and how the body handles and eliminates LY3493269 when administered orally as test compared to reference formulations in healthy participants in fed and/or fasted states. The study will also evaluate the safety and tolerability of LY3493269 in these participants. The study will last up to 43 days excluding the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants who are overtly healthy as determined by medical evaluation
* Participants with body mass index (BMI) of 19.0 to 40.0 kilograms per meter squared (kg/m²)
* Males who agree to use highly effective/effective methods of contraception and only women not of childbearing potential may participate in the trial

Exclusion Criteria:

* Have a history of atopy (severe or multiple allergic manifestations) or clinically significant multiple or severe drug allergies, or intolerance to topical corticosteroids, or severe posttreatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A dermatosis, toxic epidermal necrolysis, anaphylaxis, angioedema, or exfoliative dermatitis)
* Have a significant history of or current cardiovascular (for example, myocardial infarction, congestive heart failure, cerebrovascular accident, venous thromboembolism, etc.), respiratory, renal, gastrointestinal (GI) including involving the liver, gallbladder or gallbladder surgery, endocrine, hematological (including history of thrombocytopenia), or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk while taking the investigational product (IP); or of interfering with the interpretation of data.
* Have a mean supine heart rate (HR) less than 45 bpm or greater than 100 bpm from 2 assessments at screening.
* Have a mean supine systolic blood pressure (BP) higher than 160 mmHg and a mean supine diastolic BP higher than 95 mmHg from 2 assessments at screening
* Have undergone any form of bariatric surgery.
* Have a history of GI bleeding, or gastric or duodenal ulcers.
* Have a personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2.
* Have a history of acute or chronic pancreatitis, or elevation in serum lipase and/or amylase levels greater than 1.5 times the upper limit of normal (ULN).
* Have clinical signs or symptoms of liver disease, acute or chronic hepatitis.
* Have evidence of significant active neuropsychiatric disease as determined by the investigator.
* Have been treated with prescription drugs that promote weight loss within 3 months prior to screening.
* Are currently enrolled in a clinical study involving an IP or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have participated within the past 30 days of screening in a clinical study involving an IP; at least 5 half-lives or 30 days, whichever is longer, should have passed.
* Have an abnormality in the 12-lead electrocardiogram (ECG) at screening that, in the opinion of the investigator, increases the risks associated with participating in the study or may confound ECG (QT) data analysis, such as a QT interval corrected using Fridericia's formula (QTcF) >450 msec for males and >470 msec for females, short PR interval (<120 msec), or PR interval >220 msec, second- or third-degree atrioventricular block, intraventricular conduction delay with QRS >120 msec, right bundle branch block, left bundle branch block or Wolff-Parkinson-White syndrome.
* Have serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5x ULN or total bilirubin level (TBL) >1.5x ULN.
* Show evidence of human immunodeficiency virus infection and/or positive human immunodeficiency virus antibodies.
* Show evidence of hepatitis C and/or positive hepatitis C antibody.
* Show evidence of hepatitis B, positive hepatitis B core antibody, and/or positive hepatitis B surface antigen.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was planned to be conducted in two parts (Part A and Part B) -
  * After the completion of Part A, following a preplanned review of the safety and pharmacokinetic data from Part A, it was determined that sufficient data had been obtained. Hence, the decision was made not to proceed with Part B, and the study was terminated early.
  * Only Part A results data are reported below.
Period: Overall Study
Arm/Group | Part A: 4 mg LY3493269 Test Capsule 1 + 280 mg C10 (Fasted) | Part A: 4 mg LY3493269 Test Capsule 2 + 280 mg C10 (Fasted) | Part A: 4 mg LY3493269 Reference Tablet + 300 mg SNAC (Fasted)
Started | 12 | 15 | 15
Received at Least One Dose of Study Drug | 11 | 15 | 14
Completed | 11 | 12 | 13
Not Completed | 1 | 3 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Physician Decision | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Groups:
- Part A: 4 mg LY3493269 Test Capsule 1 + 280 mg C10 (Fasted): * Participants were administered oral doses of 4 mg LY3493269 test capsule formulation 1, co-administered with 280 mg of C10.
  * This regimen was administered once daily on Days 1, 2, and 3, following an overnight fast.
- Part A: 4 mg LY3493269 Reference Tablet + 300 mg SNAC (Fasted): * Participants were administered oral doses of 4 mg LY3493269 reference tablet formulation, co-administered with 300 mg of SNAC.
  * This regimen was administered once daily on Days 1, 2, and 3, following an overnight fast.
- Total: Total of all reporting groups
Arm/Group | Part A: 4 mg LY3493269 Test Capsule 1 + 280 mg C10 (Fasted) | Part A: 4 mg LY3493269 Test Capsule 2 + 280 mg C10 (Fasted) | Part A: 4 mg LY3493269 Reference Tablet + 300 mg SNAC (Fasted) | Total
Number analyzed (Participants) | 11 | 15 | 14 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (11.8) | 42.8 (10.4) | 39.4 (10.3) | 41.6 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2
  Male | 11 | 14 | 13 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 15 | 14 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 11 | 15 | 13 | 39
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 1 | 1
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 11 | 15 | 14 | 40

OUTCOME MEASURES:

1. Primary Outcome: Part A: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC [0-∞]) of LY3493269
Description: PK: AUC (0-∞) of LY3493269
Time Frame: Day 3: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 12, 14, 24, 48, 72,120, 288, 624 and 960 hours (h) post-dose
Population: All enrolled participants who received at least one dose of LY3493269 and had at least one evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter(ng*h/mL)
Arm/Group | Part A: 4 mg LY3493269 Test Capsule 1 + 280 mg C10 (Fasted) | Part A: 4 mg LY3493269 Test Capsule 2 + 280 mg C10 (Fasted) | Part A: 4 mg LY3493269 Reference Tablet + 300 mg SNAC (Fasted)
Number analyzed (Participants) | 11 | 15 | 14
nanograms*hours per milliliter(ng*h/mL) | 1590 (100) | 4880 (58) | 12200 (112)
Statistical Analysis 1: Comparison: Part A: 4 mg LY3493269 Test Capsule 1 + 280 mg C10 (Fasted) vs Part A: 4 mg LY3493269 Reference Tablet + 300 mg SNAC (Fasted); AUC (0-∞) was log-transformed and analyzed via mixed model for repeated measures with fixed effects for treatment, profile day and the treatment-by-day interaction, and a random effect for participant. The least square means (LSMs) and differences in LSMs were back transformed to produce the ratio between geometric least square means (GLSMs); Test type: Other; Mixed Models Analysis; Ratio of Geometric Least Squares Means = 0.130, 90% CI 2-sided [0.0741 to 0.228]
Statistical Analysis 2: Comparison: Part A: 4 mg LY3493269 Test Capsule 2 + 280 mg C10 (Fasted) vs Part A: 4 mg LY3493269 Reference Tablet + 300 mg SNAC (Fasted); AUC (0-∞) was log-transformed and analyzed via mixed model for repeated measures with fixed effects for treatment, profile day and the treatment-by-day interaction, and a random effect for participant. The LSMs and differences in LSMs were back transformed to produce the ratio between GLSMs; Test type: Other; Mixed Models Analysis; Ratio of Geometric Least Squares Means = 0.399, 90% CI 2-sided [0.237 to 0.669]

2. Primary Outcome: Part A: PK: Area Under the Concentration Versus Time Curve During One Dosing Interval (AUCτ) of LY3493269
Description: PK: AUCτ of LY3493269
Time Frame: Day 3: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 12, 14 and 24 hours (h) post-dose
Population: All enrolled participants who received at least one dose of LY3493269 and had at least one evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter(ng*h/mL)
Arm/Group | Part A: 4 mg LY3493269 Test Capsule 1 + 280 mg C10 (Fasted) | Part A: 4 mg LY3493269 Test Capsule 2 + 280 mg C10 (Fasted) | Part A: 4 mg LY3493269 Reference Tablet + 300 mg SNAC (Fasted)
Number analyzed (Participants) | 11 | 15 | 14
nanograms*hours per milliliter(ng*h/mL) | 150 (69) | 402 (66) | 1220 (108)

3. Primary Outcome: Part A: PK: Maximum Observed Drug Concentration (Cmax) of LY3493269
Description: Cmax of LY3493269
Time Frame: Day 3: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 12, 14 and 24 hours (h) post-dose
Population: All enrolled participants who received at least one dose of LY3493269 and had at least one evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part A: 4 mg LY3493269 Test Capsule 1 + 280 mg C10 (Fasted) | Part A: 4 mg LY3493269 Test Capsule 2 + 280 mg C10 (Fasted) | Part A: 4 mg LY3493269 Reference Tablet + 300 mg SNAC (Fasted)
Number analyzed (Participants) | 11 | 15 | 14
nanogram per milliliter (ng/mL) | 7.49 (80) | 25.8 (73) | 70.4 (108)
Statistical Analysis 1: Comparison: Part A: 4 mg LY3493269 Test Capsule 1 + 280 mg C10 (Fasted) vs Part A: 4 mg LY3493269 Reference Tablet + 300 mg SNAC (Fasted); Cmax was log-transformed and analyzed via mixed model for repeated measures with fixed effects for treatment, profile day and the treatment-by-day interaction, and a random effect for participant. The LSMs and differences in LSMs were back transformed to produce the ratio between GLSMs; Test type: Other; Mixed Models Analysis; Ratio of Geometric Least Squares Means = 0.106, 90% CI 2-sided [0.0620 to 0.182]
Statistical Analysis 2: Comparison: Part A: 4 mg LY3493269 Test Capsule 2 + 280 mg C10 (Fasted) vs Part A: 4 mg LY3493269 Reference Tablet + 300 mg SNAC (Fasted); [analysis description as in outcome 3, analysis 1]; Test type: Other; Mixed Models Analysis; Ratio of Geometric Least Squares Means = 0.343, 90% CI 2-sided [0.206 to 0.569]

ADVERSE EVENTS:
Time Frame: Part A: Baseline to end of follow-up (up to 43 days)
Description: All enrolled participants who received at least one dose of study drug. Participants were analyzed based on the actual treatment they received.
Arm/Group | Part A: 4 mg LY3493269 Test Capsule 1 + 280 mg C10 (Fasted) | Part A: 4 mg LY3493269 Test Capsule 2 + 280 mg C10 (Fasted) | Part A: 4 mg LY3493269 Reference Tablet + 300 mg SNAC (Fasted)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 9/11 | 11/15 | 11/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: 4 mg LY3493269 Test Capsule 1 + 280 mg C10 (Fasted) (N=11) | Part A: 4 mg LY3493269 Test Capsule 2 + 280 mg C10 (Fasted) (N=15) | Part A: 4 mg LY3493269 Reference Tablet + 300 mg SNAC (Fasted) (N=14)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — The adverse event was deemed by the investigator as not related to study treatment.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: 4 mg LY3493269 Test Capsule 1 + 280 mg C10 (Fasted) (N=11) | Part A: 4 mg LY3493269 Test Capsule 2 + 280 mg C10 (Fasted) (N=15) | Part A: 4 mg LY3493269 Reference Tablet + 300 mg SNAC (Fasted) (N=14)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (5) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Application site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Catheter site bruise (General disorders) | 1 (1) | 1 (1) | 2 (3)
Catheter site erythema (General disorders) | 2 (3) | 2 (2) | 2 (2)
Catheter site pain (General disorders) | 2 (2) | 1 (2) | 1 (1)
Catheter site phlebitis (General disorders) | 0 (0) | 0 (0) | 2 (2)
Catheter site swelling (General disorders) | 2 (2) | 2 (3) | 1 (1)
Early satiety (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hunger (General disorders) | 0 (0) | 3 (3) | 0 (0)
Medical device site erythema (General disorders) | 0 (0) | 2 (3) | 1 (1)
Medical device site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early, and Part B was not executed, as sufficient safety and pharmacokinetic data had already been obtained from Part A.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-09-18): https://cdn.clinicaltrials.gov/large-docs/43/NCT05794243/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-05): https://cdn.clinicaltrials.gov/large-docs/43/NCT05794243/SAP_001.pdf